CLINICAL TRIAL: NCT00679731
Title: A Phase 3, Multicenter, Randomized, Double-blind Study Comparing the Safety Efficacy of ABT-874 to Methotrexate in Subjects With Moderate to Severe Chronic Plaque Psoriasis
Brief Title: A Study of Safety and Efficacy Comparing ABT-874 Versus Methotrexate in Subjects With Moderate to Severe Plaque Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: M10-255; 2007-004687-47 (EudraCT Number)
Record Dates: First submitted 2008-05-15; First posted 2008-05-19 (Estimated); Last update posted 2013-01-29 (Estimated); Status verified 2013-01

CONDITIONS: Psoriasis
Keywords: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — briakinumab; Methotrexate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): ABT-874
  Interventions: Drug: ABT-874
- B (Active Comparator): Methotrexate
  Interventions: Drug: Methotrexate

INTERVENTIONS:
Drug: ABT-874 — 200 mg at week 0 and 4 and 100mg at week 8 and every 4 weeks there after administered as aSQ injection
  Arms: A
Drug: Methotrexate — 5.0 to 25 mg weekly
  Arms: B

SUMMARY:
This study is being conducted to compare the efficacy of ABT-874 versus Methotrexate in subjects with moderate to severe plaque psoriasis.

DETAILED DESCRIPTION:
This study is only being conducted in the EU and Canada

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Psoriasis for 6 MO.. BSA 10%, PASI 12 or above, PGA 3 or above

Exclusion Criteria:

* Previous exposure to anti-IL 12

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 317 (Actual)
Dates: Start 2008-04; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects who achieve a PASI 75 response relative to baseline at Week 24 | Week 24
The proportion of subjects who achieve a PGA score of 0 or 1 at Week 24 | Week 24
Proportion of subjects who achieve a PASI 75 response relative to baseline at Week 52 | Week 52
The proportion of subjects who achieve a PGA score of 0 or 1 at Week 52 | Week 52

SECONDARY OUTCOMES:
Proportion of subjects who achieve a PASI 100 response relative to baseline at Week 24 | Week 24
Changes from Baseline in the DLQI total score at Week 24 | Week 24
Proportion of subjects who achieve a PASI 100 response relative to baseline at Week 52 | Week 52
Changes from Baseline in the DLQI total score at Week 52 | Week 52

CONTACTS AND LOCATIONS:
Overall Officials: Martin Kaul, MD, Study Chair — AbbVie
Locations (43):
- Austria (3):
  - Site Reference ID/Investigator# 9904, Graz
  - Site Reference ID/Investigator# 11001, Vienna
  - Site Reference ID/Investigator# 12763, Vienna
- Site Reference ID/Investigator# 8022, Brussels, Belgium
- Canada (5):
  - Site Reference ID/Investigator# 13104, Barrie
  - Site Reference ID/Investigator# 13161, Halifax
  - Site Reference ID/Investigator# 11864, Hamilton
  - Site Reference ID/Investigator# 13223, Québec
  - Site Reference ID/Investigator# 13221, Waterloo
- Denmark (2):
  - Site Reference ID/Investigator# 11381, Aarhus
  - Site Reference ID/Investigator# 11841, Copenhagen NV
- Finland (4):
  - Site Reference ID/Investigator# 8030, Helsinki
  - Site Reference ID/Investigator# 8033, Kuopio
  - Site Reference ID/Investigator# 8021, Lahti
  - Site Reference ID/Investigator# 8026, Turku
- France (4):
  - Site Reference ID/Investigator# 11661, Créteil
  - Site Reference ID/Investigator# 11504, Nice
  - Site Reference ID/Investigator# 11161, Paris
  - Site Reference ID/Investigator# 10963, Toulouse
- Germany (7):
  - Site Reference ID/Investigator# 8025, Berlin
  - Site Reference ID/Investigator# 8024, Frankfurt am Main
  - Site Reference ID/Investigator# 8032, Hamburg
  - Site Reference ID/Investigator# 8027, Kiel
  - Site Reference ID/Investigator# 8035, Munich
  - Site Reference ID/Investigator# 8019, Münster
  - Site Reference ID/Investigator# 8023, Tübingen
- Greece (3):
  - Site Reference ID/Investigator# 13422, Athens
  - Site Reference ID/Investigator# 13462, Athens
  - Site Reference ID/Investigator# 13461, Thessaloniki
- Italy (3):
  - Site Reference ID/Investigator# 12381, Milan
  - Site Reference ID/Investigator# 9583, Modena
  - Site Reference ID/Investigator# 8551, Rome
- Netherlands (2):
  - Site Reference ID/Investigator# 11701, Amsterdam
  - Site Reference ID/Investigator# 8363, Nijmegen
- Spain (4):
  - Site Reference ID/Investigator# 13481, Barcelona
  - Site Reference ID/Investigator# 10702, Madrid
  - Site Reference ID/Investigator# 13163, Seville
  - Site Reference ID/Investigator# 8362, Valencia
- Site Reference ID/Investigator# 8185, Stockholm, Sweden
- Switzerland (2):
  - Site Reference ID/Investigator# 10203, Geneva
  - Site Reference ID/Investigator# 8020, Zurich
- United Kingdom (2):
  - Site Reference ID/Investigator# 12401, Aberdeen
  - Site Reference ID/Investigator# 8034, Manchester

REFERENCES:
- [Derived] Inzinger M, Weger W, Salmhofer W, Wolf P. Differential response of chronic plaque psoriasis to briakinumab vs. ustekinumab. Acta Derm Venereol. 2012 Jul;92(4):357-8. doi: 10.2340/00015555-1243. No abstract available. PMID 22169986
- [Derived] Reich K, Langley RG, Papp KA, Ortonne JP, Unnebrink K, Kaul M, Valdes JM. A 52-week trial comparing briakinumab with methotrexate in patients with psoriasis. N Engl J Med. 2011 Oct 27;365(17):1586-96. doi: 10.1056/NEJMoa1010858. PMID 22029980